CLINICAL TRIAL: NCT03742219
Title: Longitudinal Evaluation of Disease Prevalence in Impoverished Communities of Lima, Peru
Brief Title: Peru Longitudinal Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low level of returning participants year by year.
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, David Drozek, Associate Professor, Ohio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-X-88
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus; Hypertension; Dyslipidemias; Overweight and Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Hypertension; Dyslipidemias; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle Intervention (Experimental): Impoverished communities in Lima, Peru will be offered free medical clinics. Four communities have been chosen initially for focus over the following 10 years. These communities will be made aware of their risk for chronic lifestyle related diseases. In conjunction with the communities, specific interventions focused on a plant-based diet, physical activity, stress management and control of unhealthy habits will be devised.
  Interventions: Behavioral: Lifestyle Modification

INTERVENTIONS:
Behavioral: Lifestyle Modification — 1. Community awareness: a) individuals will be made aware of their own chronic lifestyle diseases and risk factors b) communities will be made aware of their aggregated data concerning chronic lifestyle related diseases and risk factors.
  2. Education for individuals and communities on the meaning of the lifestyle diseases and risk factors. a) individual and small group sessions explaining diseases and lifestyle measures that are helpful, b) community level education to tentatively include i) shopping guides and recipes, ii) urban gardening projects, iii) puppet shows and other community presentations, iv) literature and posters.

SUMMARY:
The purpose of this study is to evaluate the change in disease prevalence over time in impoverished urban communities in Lima, Peru.

DETAILED DESCRIPTION:
The aim is to track the changes in disease prevalence of people living in impoverished urban communities in Lima over the next 10 years.

Based on data collected in prior years and in an ongoing manner, Ohio University Global Health teams will be introducing interventions focused to positively impact disease states and trends in this population.

The current focus is on chronic lifestyle related diseases and their precursors: cardiovascular disease, hypertension, dyslipidemia, diabetes, and overweight / obesity.

ELIGIBILITY:
Inclusion Criteria:

* minors age 12-17 presenting to the free community clinic, with a responsible adult who can give consent; minors will give assent.
* consenting adults of any age who present to the clinic.

Exclusion Criteria:

* adults who are unable to give consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 861 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Weight | yearly for 10 years
  weight in kilograms will be utilized to determine body mass index
Systolic blood pressure | yearly for 10 years
  measured with a manual sphygmomanometer in millimeters of mercury
Diastolic Blood Pressure | yearly for 10 years
  measured with a manual sphygmomanometer in millimeters of mercury
glycosylated hemoglobin | periodically over 10 years
  measured in percent via fingerstick capillary blood and portable analyzer
Total cholesterol | periodically over 10 years
  measured in percent via fingerstick capillary blood and portable analyzer
Low-density lipoprotein cholesterol | periodically over 10 years
  measured in percent via fingerstick capillary blood and portable analyzer
High density lipoprotein cholesterol | periodically over 10 years
  measured in percent via fingerstick capillary blood and portable analyzer
Triglycerides | periodically over 10 years
  measured in percent via fingerstick capillary blood and portable analyzer

SECONDARY OUTCOMES:
Herth Hope Index | yearly for 10 years
  validated survey utilized to evaluate level of hope for the future
Household hunger scale | yearly for 10 years
  validated survey to measure food insecurity
Patient Health Questionnaire - 4 (PHQ-4) | yearly for 10 years
  used to evaluate depression and anxiety
Exercise vital sign | yearly for 10 years
  the minutes of exercise during the last week
Perceived Stress Scale | yearly for 10 years
  validated survey to evaluate level of stress
24 hour dietary recall | yearly for 10 years
  report of all foods consumed in the last 24 hours, which will be utilized to determine the nutritional value of dietary intake

CONTACTS AND LOCATIONS:
Overall Officials: David S Drozek, DO, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No